Conservative Management Equally Effective to New Suture Anchor Technique for Acute Mallet Finger Deformity: A Prospective Randomized Clinical Trial Date: May 23th, 2013

## **Dear Patient/ Patient's Relative**

We are conducting a scientific study. This study compares conservative treatment and internal fixation technique for mallet finger injury (tensile fracture of top of the finger). Aim of this study is conducted to determine to best treatment methods for mallet finger injury. We are planning to recruit 30 patients for study. In this study, Patients are randomized into two groups using closed opaque envelopes. One groups are treated with aluminum splint, other groups are treated with suture anchor technique. These two treatment methods have negative and positive aspects. After either treatment, you will be regularly followed up at the outpatient clinic and you will be informed of your healing progress. We will be following you up for 12 months.

There may be complications during the treatment. Should any complications occur, it will be managed by us if you wish so.

At any rate, your attendance to this study is completely up to you and you can, at any time, without being subject to any penalties or sanctions and without forfeiting any rights can deny attending the study or withdraw your consent. Your medical records before, during and after the treatment can be supervised by authorized peer councils but these records will be otherwise kept secret. Even if the results of the study are made public, your records and personal information will not.

Should any new information which may directly or indirectly affect your treatment arise during the research, you will be informed in short notice. In case of emergency, you can reach an orthopaedic consultant through 0212 414 20 00 or you may refer to our emergency department 24/7.

I have thoroughly read and reviewed the information in this consent form. I was informed about the study both in writing and verbally by the doctor named below. I am aware that I participate voluntarily and can at any time leave the study with or without an excuse.

I, without being subject to any coercion or pressure, would like to attend to the aforementioned study with my own free will.

| atients Name/Surname | | Surgery Name/Surname |
|---|---|---|
| | Date | Date |
| | Sign | Sign |
| | Patient's Relative | |
| | Date: | |
| | Sign: | |
| | L will allow just it to be used in this study mentioned above | |
| | İleride yapılması planlanan tüm araştırmalarda kullanılmasına izin veriyorum | |
| | Hicbir kosulda kullanılmasına izin vermiyorum | |